CLINICAL TRIAL: NCT01236027
Title: Collection of Biological Specimens for Development and Validation of Laboratory Procedures to Support Future Clinical Research Studies
Brief Title: Specimen Collection Study for Development and Validation of Laboratory Procedures
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Katherine Bunge, Assistant Professor, University of Pittsburgh
Other Study IDs: PRO10080337
Record Dates: First submitted 2010-11-04; First posted 2010-11-08 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Laboratory Procedure Development and Validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-negative women: HIV-negative women who agree to have specimens collected for validation of laboratory procedures
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — not applicable-no intervention

SUMMARY:
Biologic samples are necessary for development and validation of laboratory procedures (e.g. novel biological and analytical assays, explant tissue models, validation of specimen collection and transport) to support future infectious disease clinical studies. In this research study, the investigators will collect blood samples, vaginal swabs, cervical swabs, mucus/vaginal discharge, cervicovaginal lavages, vaginal and cervical biopsies, as necessary, to use in the development of laboratory processes. The investigators will obtain the sample(s) from healthy HIV negative women. Samples will be collected and sent to Magee-Womens Research Institute as laboratory specimens are needed.

ELIGIBILITY:
Inclusion Criteria:

Control Group (post-menopausal) Inclusion:

1. Females, age greater than 50 years
2. Non-pregnant
3. Post-menopausal defined as no menses or vaginal bleeding for at least 1 year
4. Agree to have HIV testing or have documentation of a negative HIV test result within the past 6 months.
5. Free from participant report and clinician observed abnormal discharge or other vaginal symptoms (with the exception of vaginal dryness) on the day of genital sample collection.
6. Willing and able to provide written informed consent.
7. Willing to provide contact information for receipt of laboratory results, as applicable.

Reproductive-aged Group Inclusion Criteria:

1. Females, 18-45 years of age
2. Non-pregnant
3. Agree to have HIV testing or have documentation of a negative HIV test result within the past 6 months.
4. Free from participant reports and clinician observed abnormal vaginal discharge or other current vaginal symptoms on the day of genital sample collection.
5. Willing and able to provide written informed consent.
6. Willing to provide contact information for receipt of laboratory results, as applicable.
7. Participant meets requirements of specific laboratory study needs (e.g. birth control method and length of use)

Exclusion Criteria:

Control Group (post-menopausal) Exclusion Criteria:

1. Use of hormone replacement therapy, including oral, vaginal and transdermal.
2. Hysterectomy.
3. An active urogenital infection within the past 14 days, including:

   1. Vaginal infections (symptomatic candidiasis, trichomonas vaginalis, and bacterial vaginosis).
   2. Cervical infections (Gonorrhea (GC), Chlamydia (CT) or mucopurulent cervicitis (MPC)).
   3. Syphilis
   4. HSV/Genital Warts
   5. Urinary Tract Infection
   6. Recent exposure to a partner with GC, CT, trichomonas, syphilis, non-gonococcal urethritis, or HIV.
4. Use of systemic or vaginal antibiotics or antifungals 14 days prior to genital sample collection.
5. Participation in a microbicide or other vaginal product study within one month of genital sample collection.
6. Use of a spermicide or spermicidally lubricated condom within one week prior to genital sample collection.
7. Use of an internal vaginal device or product with the exception of tampons within one week of genital sample collection.
8. Any other condition in the opinion of the site investigator would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data or otherwise interfere with achieving study objectives.

Reproductive-aged Group Exclusion Criteria:

1. Menopausal (including natural menopause defined as lack of menses for 12 consecutive months, in the absence of pregnancy, and surgical menopause defined as a woman who has had both ovaries removed).
2. Currently pregnant (or has been pregnant within the past 90 days) or breastfeeding
3. Hysterectomy.
4. Use of a diaphragm or NuvaRing for contraception or use of spermicide for primary contraception.
5. An active urogenital infection within the past 14 days, including:

   1. Vaginal infections (symptomatic candidiasis, Trichomonas vaginalis and bacterial vaginosis).
   2. Cervical infections (Gonorrhea (GC), Chlamydia (CT) or Mucopurulent cervicitis (MPC).
   3. Syphilis
   4. HSV/Genital Warts
   5. Urinary Tract Infection
   6. Recent exposure to a partner with GC, CT, Trichomonas, syphilis, Non-gonococcal urethritis or HIV.
6. Use of systemic or vaginal antibiotics or antifungals 14 days prior to genital sample collection.
7. Participation in a microbicide and/or contraceptive study within one month of genital sample collection.
8. Use of a spermicide or spermicidally lubricated condom within one week prior to genital sample collection.
9. Use of an internal vaginal device or product with the exception of tampons within one week of genital sample collection.
10. Any other condition in the opinion of the site investigator would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-negative women
Sampling Method: Non-Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2010-11; Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Validation of Laboratory Procedures | up to 5 years
  The primary aim of this study is to collect an adequate number of biological samples, as needed by investigators, to support development and validation of laboratory procedures necessary for upcoming topical microbicide and infectious disease research clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Hillier, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States